CLINICAL TRIAL: NCT00805090
Title: An Open-Label, Single-Dose Study to Evaluate the Safety and Pharmacokinetics of DIC075V in Subjects With Mild or Moderate Chronic Renal Insufficiency and in Subjects With Mild Chronic Hepatic Impairment Compared to Healthy Adult Volunteers and a Randomized, Open-Label, Single-Dose, Two-Way, Crossover Study to Evaluate the Safety and Pharmacokinetics of HPβCD When Administered in DIC075V Compared to Sporanox® in Healthy Adult Volunteers.
Brief Title: Open-Label, Single-Dose Study to Evaluate the Safety and PK of DIC075V in Subjects With Renal Insufficiency and Hepatic Impairment Compared to Healthy Subjects and Evaluate the Safety and Pharmacokinetics of HPβCD When Administered in DIC075V Compared to Sporanox® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Cynthia Ernst, Javelin Pharmaceuticals
Model: Crossover | Masking: None
Other Study IDs: DFC-PK-009
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Renal Insufficiency, Chronic; Hepatic Insufficiency; Healthy
Keywords: Renal; Hepatic; Healthy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatic Insufficiency | interventions — Itraconazole; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sporanox (Active Comparator): Active arm approved as an anti-fungal being used to compare HPβCD when administered in DIC075V compared to Sporanox.
  Interventions: Drug: Sporanox
- Dyloject (Experimental): Diclofenac Sodium
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Sporanox — 200 mg
  Arms: Sporanox
Drug: Diclofenac Sodium — 37.5 mg
  Arms: Dyloject

SUMMARY:
An open-label, single-dose study to evaluate the safety and pharmacokinetics of DIC075V in subjects with mild or moderate chronic renal insufficiency and in patients with mild chronic hepatic impairment compared. Additionally, the healthy adult volunteers will participate in a randomized, open-label, crossover study in which they will receive Sporanox® to compare the safety and pharmacokinetics of HPβCD when administered in DIC075V compared to Sporanox®.

DETAILED DESCRIPTION:
For the renal and hepatic subjects, following the screening visit, eligible subjects will return to the study site on Study Day 0 and remain at the site for 2 nights and 2 days. Study drug administration will occur on Study Day 1. Subjects will be discharged on Study Day 2 after the last blood sample has been collected. Subjects will return 7 ± 3 days after dosing with study drug to have final safety assessments performed. For the healthy subjects, following the screening visit, eligible subjects will return to the study site on Study Day 0 and remain at the site for 3 nights and 3 days. Study drug administration will occur on Study Day 1 and Study Day 2. Subjects will be discharged on Study Day 3 after the last blood sample has been collected. Subjects will return 7 ± 3 days after receiving the last dose of study drug to have final safety assessments performed.

ELIGIBILITY:
Inclusion Criteria (General):

* The subjects must be males or females and ≥ 18 years of age and ≤ 65 years.
* The subject must be willing and able to provide signed informed consent.
* The subject must be willing and able to stay at the clinical site for the required number of days and nights and return to the clinic in 7 ± 3 days after dosing with study drug.

Inclusion Criteria (subjects with mild or moderate chronic renal insufficiency):

* The subject must have mild or moderate chronic renal insufficiency and documented history of stable renal disease for 1 month prior to screening and clinical laboratory test results consistent with the underlying disease for renal impairment.

Inclusion Criteria (subjects with mild chronic hepatic impairment):

* The subject must have mild chronic hepatic impairment, as defined by Child-Pugh Classification A, Score of 5-6 and a bilirubin of ≤ 2.5 mg/dl.

Inclusion Criteria (for healthy subjects):

* Healthy subjects will be matched to renally impaired subjects in this study by age (+ 10 years), gender, and body weight (± 10 kg).

Exclusion Criteria:

* The subject has a known allergy or hypersensitivity to diclofenac, other NSAIDs, any of the excipients of the study preparation (hydroxypropyl-ß-cyclodextrin (HPßCD), monothioglycerol, sodium hydroxide, hydrochloric acid, and water for injection), itraconzaole or other "azole" drugs, or to any of the excipients in Sporanox (HPßCD, propylene glycol, sodium hydroxide, hydrochloric acid, or water for injection).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and pharmacokinetics of diclofenac and HPβCD following a single-dose of DIC075V in subjects with mild or moderate chronic renal insufficiency and in subjects with mild hepatic impairment compared to healthy adult volunteers. | Screening - Follow-up

SECONDARY OUTCOMES:
To evaluate the safety and pharmacokinetics of HPβCD following a single-dose of DIC075V and Sporanox in healthy adult volunteers. | Screening - Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Principal Investigator — New Orleans Clinical Center for Research; Suzanne Swann, MD, Principal Investigator — Davita Clinical Research; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Salvatore Febbraro, MD, Principal Investigator — Simbec Research
Locations (4):
- United States (3):
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota
  - New Orleans Clinical Center for Research, Knoxville, Tennessee
- Simbec Research, Ltd., Merthyr Tydfil, United Kingdom

REFERENCES:
- [Derived] Hamilton DA, Ernst CC, Kramer WG, Madden D, Lang E, Liao E, Lacouture PG, Ramaiya A, Carr DB. Pharmacokinetics of Diclofenac and Hydroxypropyl-beta-Cyclodextrin (HPbetaCD) Following Administration of Injectable HPbetaCD-Diclofenac in Subjects With Mild to Moderate Renal Insufficiency or Mild Hepatic Impairment. Clin Pharmacol Drug Dev. 2018 Feb;7(2):110-122. doi: 10.1002/cpdd.417. Epub 2017 Dec 2. PMID 29197175